CLINICAL TRIAL: NCT07203911
Title: Surgeon-performed Ultrasound for Real-time Guidance In Oral Cancer Surgeries - A Multicenter Randomized Controlled Trial
Acronym: SURGIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tobias Todsen (Other)
Collaborators: Karolinska Institutet (Other); Emory University (Other); Stanford University (Other); National Cancer Institute, Milan (Other); University of Cape Town (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor-Investigator, Tobias Todsen, MD, PhD, Ass. Prof., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p-2024-18099
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Tongue Cancer; Oral Cancer; Squamous Cell Carcinoma of the Oral Cavity or Oropharynx
MeSH Terms: conditions — Tongue Neoplasms; Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Patients will randomized to either 1)standard treatment for oral cancer 2) standard treatment for oral cancer + the use of ultrasound during surgery to guide resection process and evaluate resections margins.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Control (Active Comparator): The patients in the control group will have surgery for oral cancer conducted following the current standards for each center.
  Interventions: Other: Standard Treatment
- Intervention (Experimental): In the intervention group, surgeons will have both in-vivo and ex-vivo ultrasound at to guide the resection and evaluate surgical margins during the procedure. The in-vivo ultrasound will be employed in real-time on the tumor to guide the resection process. The surgeon begins the resection, periodically pausing to obtain real-time images of the resection plane using ultrasound. This is done by repositioning the partially resected specimen, making the resection plane visible as a hyperechoic border on the ultrasound, or by placing a small surgical instrument between the tumor/host interface to visualize the resection plane. Alternatively, the partially resected tumor can be ultrasound scanned from inside-out making the surgical margin visible nearest to the transducer. This is repeated until the tumor is completely removed.
  Interventions: Diagnostic Test: Ultrasound imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound imaging — Ultrasound will be performed during surgery in two phases: 1) in-vivo and 2) ex-vivo. In the in-vivo phase surgeons will perform intraoral ultrasound with a small intraoral transducer in order to visualize size and boundaries of tumor. Then the surgeon begins the resection periodically pausing to obtain real-time images of the resection plane and determin if resection is performed at safe distance to the tumor. In the ex-vivo phase the resected tumor will undergo ultrasound by using a motorized mechanical arm designed to hold an ultrasound transducer. This ensures standardized and reproducible scans. The purpose of the ex-vivo scan is to measure the surgical margins at the operating theatre and allow for an immediate re-resection of necessary. Surgeons in the intervention group will also have the possibility of taking biopsies for frozen section analyses.
  Arms: Intervention
Other: Standard Treatment — Standard surgical treatment of oral cancer
  Arms: Control

SUMMARY:
The goal of this clinical trial is to improve the surgical treatment of patients with oral cancer. We will explore whether the use of surgeon performed ultrasound during these surgeries result in better tumor removal. We hypothesize that using intraoperative ultrasound to assist the resection results in more frequent clear surgical margins in oral cancer surgeries compared to standard methods. This improvement is associated with a reduced need for post-operative adjuvant therapies such as radiotherapy and reoperation, lower mortality rates, lower cancer recurrence, and enhanced quality of life for patients undergoing surgery for oral cancer.

Participants will be randomized to either the control or intervention group:

* Control group will receive standard treatment for oral cancer.
* Intervention group will in addition to the standard treatment have surgery performed using ultrasound to guide the resection and evaluate resection margins intraoperatively.

Outcomes:

* Number of free surgical margins between control and intervention group.
* Intraoperative surgeon assessed surgical margins compared to final histology report.
* Dysphagia and quality of life questionnaires.
* Recurrence rates.
* Mortality rates.

All participant will be followed-up at 3 months and 12 months with:

* MDADI dysphagia questionnaire
* EORTC head and neck cancer quality of life questionnaire
* Follow-up on recurrrence and mortality.

DETAILED DESCRIPTION:
Background:

Surgery is the primary treatment for early-stage oral cancer, aiming to completely remove the tumor along with a margin of healthy tissue to ensure a clear surgical margin. However, in up to 50% of cases, the tumor is not entirely removed, leading to higher rates of cancer recurrence and mortality. This challenge often arises from difficulty distinguishing tumor tissue from healthy tissue during the operation. Studies have shown that ultrasound can effectively make this distinction. This project investigates using B-mode in-vivo and ex-vivo ultrasound to assist surgeons in the resection of the tumor. The objective is to enhance accuracy during these surgeries by use of ultrasound. Consequently, we hope to minimize the need for adjuvant therapies, potentially enhancing patients' quality of life and reducing cancer recurrence and mortality rates.

Study population:

Inclusion criteria

• Patients scheduled for surgical treatment of biopsy-proven T1-T3 oral squamous cell carcinoma.

Exclusion criteria

* Age < 18 years.
* Oral cancer with suspected bone involvement.
* Unable to understand verbal or written information.
* Prior radiotherapy treatment of oral cavity cancer.
* Tumor not visible on ultrasound.

Methods:

We plan to conduct a multicenter randomized controlled trial at seven otorhinolaryngology-Head and Neck Surgery departments in Europe, USA and Africa. The trial is anchored in Rigshospitalet, Copenhagen (Denmark).

Patients who meet the study´s criteria will be assigned either the control - or intervention group.

* Patients in the control group will have surgery for oral cancer conducted following the current standards for each center. The oral cancer tumor will be excised without having an ultrasound machine available to guide the resection. Then, the surgeon will take additional biopsies either from the in-vivo wound edges or from the specimen depending on local guidelines. Then the biopsies will be sent to the pathology department for frozen-section analysis. The surgeon might revise the resection or terminate the operation based on the frozen-section result. If the frozen-section analysis indicates an inadequate margin, the surgeon will, if possible, excise additional tissue from the wound, and the measured margin will be adjusted accordingly.
* In the intervention group, surgeons will have both in-vivo and ex-vivo ultrasound at their disposal to guide the resection and evaluate surgical margins during the procedure. The in-vivo ultrasound will be employed in real-time on the tumor to guide the resection process. Initially, tumor dimensions are measured using a Fujifilm robotic ultrasound probe or a hockey stick probe, and a 10 mm margin is marked from the tumor's boundaries. The surgeon begins the resection, periodically pausing to obtain real-time images of the resection plane. This is done by repositioning the partially resected specimen, making the resection plane visible as a hyperechoic border on the ultrasound, or by placing a small surgical instrument between the tumor/host interface to visualize the resection plane. Alternatively, the partially resected tumor can be ultrasound scanned from inside-out making the surgical margin visible nearest to the transducer. This is repeated until the tumor is completely removed.

After tumor removal, the specimen will undergo an ex-vivo ultrasound scan. In this phase, we will use a motorized mechanical transducer holder to hold the transducer to obtain standardized and reproducible B-mode cross-sectional images of the resected tissue allowing for margin measurement in the operating room. This imaging along with the margin measurements will help surgeons decide whether to perform an immediate re-resection or to conclude the operation. The use of ultrasound will not replace standard procedures, but should instead be viewed as an add-on tool. Therefore, surgeons in the intervention group will have the possibility to take biopsies for frozen section analyses.

ELIGIBILITY:
Inclusion criteria

• Patients scheduled for surgical treatment of biopsy-proven T1-T3 oral squamous cell carcinoma.

Exclusion criteria

* Age < 18 years.
* Oral cancer with suspected bone involvement.
* Unable to understand verbal or written information.
* Prior radiotherapy treatment of oral cavity cancer.
* Tumor not visible on ultrasound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Free surgical margin | 2 weeks.
  Free surgical margin defined as resection margin above 5mm on final histopathology report. Reported as dichotomous variable "free surgical margin yes/no"

SECONDARY OUTCOMES:
Surgeon assessed margins | 2 weeks.
  Surgeons will intraoperatively try to predict the surgical margin on final histopathology report. This is important as it is not always possible to obtain free margin (above 5 mm). Therefore, this outcome will explore whether ultrasound is a viable tool to assess surgical margins regardless of whether the surgeon has obtained a "free surgical margin".
Dysphagia questionnaire | 12 months
  MD Anderson Dysphagia Inventory to assess dysphagia at 3 and 12 months.
Cancer recurrence | 24 months
  This outcome will explore whether the use of ultrasound leads to more complete removal of cancerous tissue.
Survial | 24 months
  This outcome will explore whether an expected increased frequency of "free surgical margins" in the intervention group also reflects on survival.
Quality of life questionnaire | 12 months
  EORTC HN43 quality of life questionnaire in order to assess quality of life after head and neck cancer.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (2):
  - Stanford Otolaryngology - Head & Neck Surgery Department, Stanford, California
  - Emory University Hospital, Atlanta, Georgia
- Denmark (2):
  - Department of Otorhinolaryngology Head and Neck Surgery, Aarhus
  - Department of Otorhinolaryngology Head and Neck Surgery and Audiology, Rigshospitalet, Copenhagen
- Istituto Nazionale Tumori of Milan, Milan, Italy
- Groote Schuur, Cape Town, South Africa
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in surgical treatment of oral cancer. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact daniel.julius.lauritzen@regionh.dk